CLINICAL TRIAL: NCT01164943
Title: Aneuploidy Rate Impact in Oocyte From Egg Donation Cycle With Different Stimulation Protocol: Recombinant FSH vs Human FSH
Brief Title: Aneuploidy Rate and Stimulation Protocol: Recombinant Follicle Stimulating Hormone (FSH) Versus Human FSH
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: IVI Madrid (Other)
Responsible Party: Principal Investigator, Juan A Garcia-Velasco, PhD, MD, IVI Madrid
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MAD-FB-04-2010-01
Record Dates: First submitted 2010-07-16; First posted 2010-07-19 (Estimated); Last update posted 2016-02-25 (Estimated); Status verified 2015-04

CONDITIONS: Aneuploidy Rate
MeSH Terms: interventions — Follicle Stimulating Hormone, Human

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Human FSH (Active Comparator)
  Interventions: Procedure: Stimulation with human FSH
- Recombinant FSH (Active Comparator)
  Interventions: Procedure: Stimulation with recombinant FSH

INTERVENTIONS:
Procedure: Stimulation with human FSH — Human FSH
  Arms: Human FSH
Procedure: Stimulation with recombinant FSH — Recombinant FSH
  Arms: Recombinant FSH

SUMMARY:
Several stimulation protocols have been used in in vitro fertilization (IVF) in a cycle of egg donation; recombinant FSH and human FSH are included. The effect of each kind of hormone on aneuploidy rate it is unknown. If there was an increase on aneuploidy rate of one of these stimulation protocols, there will be a negative effect on the successful rates in the egg donation cycles. The aim of this study is to observe if there is a different in aneuploidy rate and morphological oocyte parameters between different stimulation protocols.

ELIGIBILITY:
Inclusion Criteria:

* Egg donation cycles with more than 8MII in oocyte retrieval day

Exclusion Criteria:

* Male factor
* Uterine malformations
* genetic alterations

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2010-07; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Aneuploidy Rate | 2011 January
  Analysis of all nuclei fixed

SECONDARY OUTCOMES:
Oocyte morphology | 2011 january
  Analysis of all oocytes
Outcome rates (implantation, pregnancy and miscarriage rate) | 2011 April
  Time requierd to know all the implantation, pregnancy and miscarriage rate

CONTACTS AND LOCATIONS:
Locations (1):
- Insituto Valenciano de Infertilida, Spain, Madrid, Madrid, Madrid, Spain